STATURE: A prospective observational study of the relation  $\underline{S}$  hip be  $\underline{T}$  ween or  $\underline{A}$ I DM $\underline{T}$  b  $\underline{UR}$  den and adh  $\underline{E}$  rence in people with MS.

NCT: TBC

13/07/2020

## **Online Participant Consent Process**

Following provision of the information statement and contact with a member of the STATURE research team, who will ask the potential participant if they would like them to talk through the salient points of the information statement and provide them an opportunity to ask questions, interested potential participants will be emailed a link to provide online study consent before completing the baseline survey.

The provided link will take participants to the introduction page of online process and explain that they will be requested to provide consent to the research and then undertake the first survey. Participants will press **NEXT** to continue or **CANCEL** to abort.

The second page will provide the consent form:

## **Consent Form**

**Title** STATURE: A prospective observational study of the relationShip

be<u>T</u>ween or<u>Al DMT</u> b<u>UR</u>den and adh<u>E</u>rence in people with MS.

Short Title STATURE: Relationship Between Oral Disease Modifying

Treatment Burden and Adherence in MS

**Protocol Number** 

Project Sponsor

Coordinating Principal

Investigator/

Monash University

Ass. Prof. Ernest Butler Dr Lisa Grech, Ms Michelle Allan

Associate Investigator(s)

Mr Tim O'Maley, Ms Sharryn Savickas, Ms Meena Sharma, Mr

Paul Stockle, Ms Adriana Cartwright

**Location** Remote

## **Declaration by Participant**

I **[insert full name]** have read the Participant Information Sheet or someone has read it to me in a language that I understand.

I understand the purposes, procedures and risks of the research described in the project.

I have had an opportunity to ask questions and I am satisfied with the answers I have received.

I freely agree to participate in this research project as described and understand that I am free to withdraw at any time during the project without affecting my future healthcare.

| ☐ Yes I consent to participation in this research project. |
|---|
| ☐ Cancel, I have decided not to participate. |
| If they tick Yes a popup screen will appear stating: |
| You have agreed to participate in the research project "STATURE: Relationship Between Oral DMT Burden and Adherence in MS". This includes undertaking three questionnaires (the first now, one in 3-months and one 12-months) and allowing secure and confidential access to study related medical records and Medicare information. Do you understand? |
| □ Cancel |
| If they tick Cancel (at either of the above points) this will take potential participant to a screen stating: |
| Thank you for your consideration in this research. Your decision not to participate will not affect |

If the participant ticks Yes to the popup screen, they will then be taken to the next screen to commence the questionnaire.

your relationship with healthcare providers and any associated services in any way.